CLINICAL TRIAL: NCT02892045
Title: Sensitivity and Specificity of the New Mindray 3-Directional Neuromuscular Transmission Module Versus the Relaxometer Mechanomyograph and Versus TOF-Watch Acceleromyograph for Neuromuscular Block Monitoring
Brief Title: Mindray Neuromuscular Transmission Transducer
Acronym: NMT1
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Collaborators: Dalian Medical University (Other)
Responsible Party: Principal Investigator, Ashraf Dahaba, MD, Principal Investigator, Suez Canal University
Other Study IDs: NMT1
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular block; monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MMG versus Mindray NMT: 24 patients where Mindray NMT is monitoring one hand versus Mechanomyograph on the other hand accessible in supine position, alternately right and left hands monitoring neuromuscular block of rocuronium neuromuscular blocking agent 0.6 mg/kg.
  Interventions: Device: MMG
- TOFWatch versus Mindray NMT: 24 patients where Mindray NMT is monitoring one hand versus TOF-Watch Acceleromyograph on the other hand accessible in supine position, alternately right and left hands monitoring neuromuscular block of rocuronium neuromuscular blocking agent 0.6 mg/kg

INTERVENTIONS:
Device: MMG — neuromuscular monitoring device
  Groups: MMG versus Mindray NMT

SUMMARY:
A new NMT module from Mindray (Mindray Co. Shenzhen, People's Republic of China.) claims to measure 3 directional accelerography. The aim of the study is to compare the neuromuscular block of rocuronium 0.6 mg/kg (twice the 95% effective dose, ED95) monitored by the NMT versus that monitored by the Relaxometer Mechanomyograph on the other hand in Group 1, and versus the TOF-Watch on the other hand in Group 2 to clinically evaluate the new system for its diagnostic accuracy.

DETAILED DESCRIPTION:
Mechanomyography (MMG) is regarded as the standard method for precise quantification of neuromuscular block. The conventional MMG measures the exact force of muscle contraction in response to electric stimulation of the ulnar nerve. MMG quantifies the neuromuscular function by measurement of the force displacement. However the equipment is rather bulky, takes time to set up, requires a rigid support of the arm in an often-crowded operating room. This limits its clinical use in the daily anesthesia practice. Acceleromyography is based on the acceleration of a piezo-electrode. A new NMT module from (Shenzhen, People's Republic of China.) claims to measure 3 directional accelerography. The aim of the study is to compare the neuromuscular block of rocuronium 0.6 mg/kg (twice the 95% effective dose, ED95) monitored by the NMT to that monitored by the Relaxometer Mechanomyograph in Group 1, and versus TOF-Watch Acceleromyograph in Group 2 to clinically evaluate the new system for its diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 24 patients with Mindray NMT monitoring on one hand versus MMG Mechanomyograph on the other hand in Group 1 with both hands accessible in supine position alternately right and left hands monitoring neuromuscular block of rocuronium neuromuscular blocking agent 0.6 mg/kg
* 24 patients with Mindray NMT monitoring one hand versus TOF-Watch Acceleromyograph on the other hand in Group 2 with both hands accessible in supine position alternately right and left hands monitoring neuromuscular block of rocuronium neuromuscular blocking agent 0.6 mg/kg.

Exclusion Criteria:

* Both hand inaccessible in supine position, patients receiving drugs interfering with rocuronium neuromuscular block, or patients with small joint arthritis that could affect neuromuscular monitoring.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 48 patients as follows 24 patients with Mindray NMT monitoring one hand versus Mechanomyograph on the other hand in Group 1, and 24 patients with Mindray NMT monitoring one hand versus TOF-Watch Acceleromyograph on the other hand in Group 2 with hands in both Groups accessible in supine position, alternately right and left hands monitoring neuromuscular block of rocuronium neuromuscular blocking agent 0.6 mg/kg.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics parameters (onset time 95% maximum depression, clinical duration T1 25%, and full recovery 0.8-0.9 TOF ratio neuromuscular block | one year
  this will determine the Sensitivity and specificity versus MMG mechanomyography

SECONDARY OUTCOMES:
Bland and Altman bias and limits of agreement | one year
  Bias is difference between the 2 monitors and the limits of agreement is bias +/- 1.96 SD.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Dahaba, MD, Principal Investigator — Suez Canal University
Locations (2):
- Sarajevo medical University, Sarajevo, Bosnia and Herzegovina
- Dalian Medical University, Dalian, Dalian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Viby-Mogensen J, Engbaek J, Eriksson LI, Gramstad L, Jensen E, Jensen FS, Koscielniak-Nielsen Z, Skovgaard LT, Ostergaard D. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents. Acta Anaesthesiol Scand. 1996 Jan;40(1):59-74. doi: 10.1111/j.1399-6576.1996.tb04389.x. PMID 8904261